CLINICAL TRIAL: NCT04867629
Title: No Evidence of Impact of Seed Oil Intake on Biomarkers of Coronary Artery Disease, Chronic Kidney Disease and Diabetes in Healthy Adults With Overweight and Obesity - Result From a Blinded Randomised Control Trial
Brief Title: Impact of Rapeseed and Sunflower Oils on Proteomic Biomarkers of Diseases.
Acronym: DOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Emilie Combet, Senior lecturer, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DOC
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Diseases
Keywords: rapeseed oil; sunflower oil; proteomics; cardiometabolic; cardiovascular; fatty acids; monounsaturated fatty acids; seed oils; dietary fat
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Rapeseed Oil; Sunflower Oil

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Investigator
Masking Description: Oils were in identical amber glass bottles labelled A or B. Oils blinded to participants and investigators. However, the control group was unblinded due to them not receiving any intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rapeseed oil (Experimental): Participants asked to consume 20mL of rapeseed oil raw every day for 12 weeks
  Interventions: Dietary Supplement: Rapeseed oil
- Sunflower oil (Active Comparator): Participants asked to consume 20mL of sunflower oil raw every day for 12 weeks
  Interventions: Dietary Supplement: Sunflower oil
- Habitual diet (No Intervention): Participants asked to maintain their habitual diet for 12 weeks

INTERVENTIONS:
Dietary Supplement: Rapeseed oil — 20mL of rapeseed oil to be consumed daily in replacement to habitual oil
  Other Names: RO
  Arms: Rapeseed oil
Dietary Supplement: Sunflower oil — 20mL of sunflower oil to be consumed daily in replacement to habitual oil
  Other Names: SO
  Arms: Sunflower oil

SUMMARY:
This study will test the impact of vegetable oils with contrasting fatty acids composition on biomarkers of health (cardiovascular, kidney diseases and diabetes) after twelve weeks supplementation. We will use sunflower oil (high in PUFAs), rapeseed oil (high in MUFAs, locally produced) and a non-intervention control. We have developed a sensitive and selective urinary proteomic biomarker of cardiovascular disease which we will use in a double-blinded randomised study.

DETAILED DESCRIPTION:
The intervention follows a parallel double-blind randomised control design. The intervention duration is 12 weeks, with a mid-point assessment at 6 weeks. Randomisation to groups; rapeseed oil, sunflower oil or habitual diet is performed using a block stratified allocation based on age (under or over 45) and BMI (under or over 30kg/m2) and is carried out remotely via phone.

Participants allocated to either oil groups are instructed to consume the oils uncooked, as a partial replacement to their habitual fat intake. Participants in the control group are asked to not change any aspect of their diet.

Spot urine samples are collected from all participants at all time points for measurement of the primary outcome (proteomic biomarker score). Urine is collected in a plastic tube, mid-flow, as the second urination of the day at baseline, 6 and 12 weeks.

Fasting venous blood is collected for the assessment of secondary outcomes, at baseline, 6 weeks and 12 weeks. Participants are also asked to complete a 2-day food diary at weeks 0, 6 and 12

ELIGIBILITY:
Inclusion Criteria:

* Overweight adults with a BMI>25 and/or a large waist (Male >102cm and female >88cm),
* Aged 25-75 years
* No history of chronic disease of the GI tract
* Not taking medication (other than the contraceptive pill).

Exclusion Criteria:

* Pregnant or lactating
* Allergy to any vegetable oils and vegetable oil-derived products

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Proteomic biomarkers | 0, 6, 12 weeks
  Changes in proteomic biomarker scores of coronary artery disease (CAD238), chronic kidney disease (CKD273)

SECONDARY OUTCOMES:
Blood lipids | 0, 6, 12 weeks
  Changes in concentrations of plasma glucose, triglycerides, total cholesterol, high density lipoprotein,
Inflammation markers | 0, 6, 12 weeks
  Changes in concentrations of plasma interleukin 6, tumor necrosis factor, matrix metallopeptidase 9
Oxidative stress biomarkers | 0, 6, 12 weeks
  Changes in concentrations of plasma fructosamine, AGE, RAGE

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicol K, Mansoorian B, Latosinska A, Koutroulaki A, Mullen B, Combet E. No evidence of differential impact of sunflower and rapeseed oil on biomarkers of coronary artery disease or chronic kidney disease in healthy adults with overweight and obesity: result from a randomised control trial. Eur J Nutr. 2022 Sep;61(6):3119-3133. doi: 10.1007/s00394-022-02810-5. Epub 2022 Apr 5. PMID 35381848